CLINICAL TRIAL: NCT00170547
Title: Immunogenicity and Safety of a Split, Inactivated, Trivalent Influenza Vaccine Administered by Intradermal Route Compared to an Intramuscular Vaccination With Fluzone(R) in Healthy Adults
Brief Title: Comparison of Delivery Routes of Flu Vaccine in Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 05-0075
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2006-07

CONDITIONS: Influenza
Keywords: inactivated, trivalent, influenza, vaccine, Fluzone
MeSH Terms: conditions — Influenza, Human

ARMS (4):
- Group 3 (Experimental): 382 subjects will receive one 3 mcg dose of Fluzone intradermally using the Mantoux technique on Day 0,
  Interventions: Biological: Trivalent inactivated influenza vaccine
- Group 4 (Experimental): 382 subjects will receive one 15 mcg dose Fluzone vaccine intramuscularly (IM) on Day 0,
  Interventions: Biological: Trivalent inactivated influenza vaccine
- Group 1 (Experimental): 382 subjects will receive one 6 mcg dose of Trivalent inactivated influenza vaccine (TIV) intradermally (ID) with the BD ID System on Day 0,
  Interventions: Biological: Trivalent inactivated influenza vaccine
- Group 2 (Experimental): 382 subjects will receive one 9 mcg dose of TIV intradermally (ID) with the BD ID System on Day 0,
  Interventions: Biological: Trivalent inactivated influenza vaccine

INTERVENTIONS:
Biological: Trivalent inactivated influenza vaccine — A synthetic vaccine consisting of three inactivated influenza viruses: two different influenza type A strains and one influenza type B strain.. Group 4: 382 subjects receive Fluzone 15 mcg IM on day 0
  Arms: Group 4
Biological: Trivalent inactivated influenza vaccine — A synthetic vaccine consisting of three inactivated influenza viruses: two different influenza type A strains and one influenza type B strain. Group 1: 382 subjects receive 6 mcg ID with BD system. Group 2: 382 subjects receive 9 mcg ID with BD system, all doses on day 0.
  Arms: Group 1; Group 2
Biological: Trivalent inactivated influenza vaccine — A synthetic vaccine consisting of three inactivated influenza viruses: two different influenza type A strains and one influenza type B strain..Group 3: 382 subjects receive 3 mcg Fluzone ID using Mantoux technique on day 0.
  Arms: Group 3

SUMMARY:
This protocol is to compare the immune response of different influenza vaccines given by two different routes of administration in healthy adults ages 18 to 64 years.

DETAILED DESCRIPTION:
This is a multi-center, randomized, partially blinded trial to compare the safety and immunogenicity of intramuscularly versus intradermally administered influenza vaccine in healthy 18-64 year old adults. Subjects will have blood drawn immediately prior to and approximately three to four weeks after vaccination. After the completion of the trial, all subjects will be offered influenza vaccine of the 2005-2006 formulation.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is healthy, as determined by medical history
2. Over 18 years of age and not yet 65 years old
3. Provides written informed consent
4. Able to attend all scheduled visits and to comply with all trial procedures
5. Women may be menopausal of 1 year or more or sugically sterile. Women of child-bearing potential must agree to be abstinent or to use a licensed form of barrier or hormonal contraception for the entire study period, and have a negative pregnancy test within 24 hours prior to vaccination.

Exclusion Criteria:

1. Breast-feeding
2. Receipt of an investigational drug, biologic or device in the 4 weeks preceding the trial vaccination
3. Planned participation in another clinical trial during the present trial period
4. History of Guillain-Barré Syndrome
5. Congenital or acquired immunodeficiency, immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months, or long-term systemic corticosteroid therapy
6. Hypersensitivity to any of the vaccine components (including eggs or egg products or thimerosol and gelatin) or history of a life-threatening reaction to the trial vaccine or a vaccine containing the same substances
7. Chronic illness that could interfere with trial conduct or completion
8. Blood or blood-derived products received in the past 3 months
9. Has received any inactivated vaccine within 2 weeks or live vaccine within 4 weeks prior to enrollment into this study
10. Vaccination planned within the 4 weeks following the trial vaccination
11. Known current HIV, hepatitis B (HBsAg) or hepatitis C infection or seropositivity
12. Prior vaccination against influenza within the past 6 months
13. Allergy shot in the 7-day period prior to enrollment and must not be scheduled to receive any allergy shots in the 7-day period after enrollment
14. On coumadin or heparin therapy or has known thrombocytopenia or bleeding disorder contraindicating vaccination
15. Subject deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized without his/her consent
16. Febrile illness temperature >= 37.5°C on Day 0, prior to enrollment and vaccination
17. Any condition, that, in the opinion of the investigator, would pose a health risk to the participant
18. History of alcohol or drug abuse in the last 5 years
19. Planned travel outside the US between vaccination and the second study visit
20. Presence of any active skin disease at the injection site that, in the opinion of the Investigator, would impact vaccine delivery or assessment of vaccination site

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1597 (Actual)
Dates: Start 2005-09; Primary Completion 2006-01 (Actual); Study Completion 2006-02

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Stanford University School of Medicine, Stanford, California
  - UCLA Center For Vaccine Research, Torrance, California
  - University of Iowa - Vaccine Research & Education Unit, Iowa City, Iowa
  - University of Maryland Baltimore, Baltimore, Maryland
  - Saint Louis University, St Louis, Missouri
  - University of Rochester Medical Center - Strong Memorial Hospital - Infectious Diseases, Rochester, New York
  - Duke Health Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Vanderbilt University, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas